CLINICAL TRIAL: NCT06827080
Title: Study on the Safety, Tolerability, and Preliminary Efficacy of 161Tb-NYM032 in Patients with Metastatic Castration-Resistant Prostate Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhengguo Chen (Other)
Responsible Party: Sponsor-Investigator, Zhengguo Chen, Chief Physician, Mianyang Central Hospital
Organization: Mianyang Central Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MianyangNC
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Castration-resistant Prostate Cancer, MCRPC; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 161Tb-NY032 (Experimental)
  Interventions: Drug: 30 mCi NYMO32; Drug: 50 mCi NYMO32; Drug: 80 mCi NYMO32; Drug: 130 mCi NYMO32; Drug: 200 mCi NYMO32

INTERVENTIONS:
Drug: 30 mCi NYMO32 — The initial dose is set at 30 mCi.
Drug: 50 mCi NYMO32 — The dose will be escalated to 50 mCi.
Drug: 80 mCi NYMO32 — The dose will be escalated to 80 mCi.
Drug: 130 mCi NYMO32 — The dose will be escalated to 130 mCi.
Drug: 200 mCi NYMO32 — The maximum dose is set at 200 mCi.

SUMMARY:
161Tb-NYM032 is a radiopharmaceutical labeled with a PSMA ligand, used for the treatment of metastatic castration-resistant prostate cancer, which is needed for clinical trial to be conducted.

ELIGIBILITY:
**1. Inclusion Criteria**

1. The participant voluntarily signs the informed consent form and is able to complete the trial according to the protocol requirements.
2. Male, aged 18 years or older.
3. Diagnosed with metastatic castration-resistant prostate cancer (mCRPC) as per PCWG3 criteria.
4. Positive results on 68Ga-NYM032 positron emission tomography (PET)/computed tomography (CT) scan.
5. Must have received at least one NAAD treatment (e.g., enzalutamide and/or abiraterone) or at least one taxane-based treatment regimen, or be intolerant to or refuse taxane therapy for metastatic castration-resistant prostate cancer.
6. ECOG performance status of 0-2.
7. Expected survival of ≥6 months.
8. Laboratory parameters must meet the following:

   1. ALT and AST must not exceed 3 times the upper limit of normal (ULN); BUN and Cr must not exceed 1.5 times the ULN.
   2. Blood counts: WBC ≥3.5×10^9/L, PLT ≥100×10^9/L, Hb ≥90 g/L.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-11 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
PSA | 5-6 weeks after each administration.
  PSA levels can be used to monitor the treatment efficacy, disease progression, or recurrence of prostate cancer. A decrease in PSA levels after treatment usually indicates effective therapy, while an increase in PSA levels may suggest disease recurrence or progression.
68Ga-NYM032 PET/CT | **5-6 weeks after the second and fourth administrations in the same dose-escalation cohort.**
  **Reflect the PSMA expression level in the patient's lesions.**

IPD SHARING:
Plan to Share IPD: Undecided